CLINICAL TRIAL: NCT06095843
Title: "Bony Changes Around Dental Implant Placed in Free Vascularized Fibular Graft Versus Non-Vascularized Iliac Crest Graft in Mandibular Reconstruction"
Brief Title: "Bony Changes Around Dental Implant in Free Fibular Graft Versus Non-Vascularized Iliac Crest Graft"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Maged Mohamed Mostafa, Assistant lecturer of oral and maxillofacial surgery, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9D
Record Dates: First submitted 2022-11-08; First posted 2023-10-23 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Crestal Bone Loss; Survival Rate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- implants in free vascularized fibular flap (Active Comparator): placement of dental implants in free fibular flaps after mandibular reconstruction
  Interventions: Procedure: placement of dental implants
- implants in non-vascularized iliac crest grafts (Active Comparator): placement of dental implants in non-vascularized iliac crest grafts after mandibular reconstruction
  Interventions: Procedure: placement of dental implants

INTERVENTIONS:
Procedure: placement of dental implants — placement of dental implants in mandibular reconstruction.

SUMMARY:
The goal of this clinical trial is to evaluate the bony changes around dental implants in non-vascularized iliac crest grafts and free vascularized fibular flap in mandibular reconstruction.

The main question it aims to answer are:

• evaluate the bony changes around dental implants and it's survival rate in both groups

DETAILED DESCRIPTION:
The current prospective study was conducted on 10 patients that were selected and admitted for early or delayed mandibular reconstructive surgery from the outpatient who were referred to the department of Oral and Maxillofacial Surgery Faculty of Dentisry, Ain Shams University in the period from January 2018 till June 2022.

The patients in this study were divided into two groups. First group endured non-vascularized iliac crest grafting with delayed implant insertion while the second group endured vascularized fibular flap with delayed implant insertion. Implant placement was done six months after performing reconstructive surgery.At the second stage surgery, all succeeded implants were loaded with fixed implant supported prothesis. Follow- up was done 1 week, 2 weeks, 4 weeks, 8 weeks and 12 weeks postoperatively.

Crestal bone stability was analyzed using CBCT radiographs along with the percentages of of the survived implants and ISQ values were measured using an ostell device.

ELIGIBILITY:
Inclusion Criteria:

* patients following traumatic injuries
* gunshot injuries
* tumor ablative surgeries
* osteomylitis and osteonecrosis affecting the mandible

Exclusion Criteria:

* cardiovascular or pulmonary disease
* vascular or bone disorder
* previous fractures or surgeries related to the donor site

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
bony changes around dental implants | 1 year
  measuring crestal bone loss (mm)
survival rate of dental implants | 1 year
  measuring survival rate of dental implants (%)
stability of dental implants | 1 year
  measuring primary and secondary stability (ISK)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No